CLINICAL TRIAL: NCT03241979
Title: The Effects of Transnasal Humidified Rapid Insufflation Ventilator Exchange (THRIVE) on the Oxygenation in Pediatric Patients Under Tubeless Airway Surgery - a Physiologic Study
Brief Title: THRIVE in Pediatric Laryngeal Microsurgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Other Study IDs: H1706-204-866
Record Dates: First submitted 2017-07-28; First posted 2017-08-08 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Laryngoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- laryngeal microsurgery

SUMMARY:
Transnasal High-flow rapid-insufflation ventilatory exchange (THRIVE) has been shown to benefit oxygenation, ventilation and upper airway patency in a range of clinical scenarios, however its use in spontaneously breathing pediatric patients undergoing tubeless airway surgery has not been described. This is a physiologic study that evaluates the feasibility of THRIVE during pediatric airway surgery under self-respiration.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing laryngeal microsurgery with spontaneous ventilation

Exclusion Criteria:

* Severe gastrointestinal reflux disease Neuromuscular disease Central hypoventilation

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
number of low saturation events | Intraoperative
  oxygen saturation decrease lower than 90%

CONTACTS AND LOCATIONS:
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim EH, Ji SH, Lee JH, Kim JT, Jang YE, Kwon SK, Kim HS. Use of high-flow nasal oxygen in spontaneously breathing pediatric patients undergoing tubeless airway surgery: A prospective observational study. Medicine (Baltimore). 2022 Jul 8;101(27):e29520. doi: 10.1097/MD.0000000000029520. PMID 35801795